CLINICAL TRIAL: NCT01407042
Title: Patellofemoral Pain After Unicondylar Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Michael Liebensteiner, MD, PhD, Medical University Innsbruck
Other Study IDs: PFJ-UKA-1
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Mobile-bearing Unicondylar Knee Arthroplasty
Keywords: unicondylar knee arthroplasty; mobile-bearing; patellofemoral pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- mb-UKA: Patients with unicondylar osteoarthritis of the knee
  Interventions: Procedure: mobile-bearing unicondylar knee arthroplasty

INTERVENTIONS:
Procedure: mobile-bearing unicondylar knee arthroplasty — mobile-bearing unicondylar knee arthroplasty

SUMMARY:
Unicondylar knee arthroplasty (UKA) is a proven procedure in patients suffering from unicompartmental knee osteoarthritis. Two different types of UKA design are available - both with different pros and cons. The so-called 'mobile-bearing UKA' requires the removal of an additional amount of cartilage and bone close to the implantat. It is unclear whether this is of clinical relevance.

We speculate that the amount of cartilage/bone removal is related to the clinical outcome of the UKA-surgery.

In patients receiving a mobile-bearing UKA that amount of cartilage/bone removal is measured during the surgery. The clinical success of the procedure will be determined with certain knee questionnaires (Kujala & KOOS)preoperatively, 3 months postoperatively, 6 months postoperatively and 1 year postoperatively. Additionally, the so-called bone-remodelling around that area of resected cartilage and bone will be measured (SPECT-CT) postoperatively.

The three variables (removed amount of cartilage/bone; clinical success with regard to the questionnaires; bone remodelling) are then analyzed with statistical methods to find out potential assoziations among them.

ELIGIBILITY:
Inclusion Criteria:

- osteoarthritis or osteonecrosis in the medial or lateral tibiofemoral compartment

Exclusion Criteria:

* failed upper tibial osteotomy
* insufficiency of the collateral or anterior cruciate ligaments
* a fixed varus or valgus deformity (not passively correctable) above 15°
* a flexion deformity greater than 15°
* rheumatoid arthritis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients scheduled for unicondylar knee arthroplasty at the Dept. for orthopaedic surgery of our medical university
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Size of anterior femoral notch | day 0
  Required cartilage / bone removal adjacent to the femoral implant
Kujala Score changes | -1 days, 3 months, 6 months, 1 year
KOOS questionnaire changes | -1 days, 3 months, 6 months, 1 year
Radionuclide tracer uptake at the surgically created notch | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Innsbruck Medical University, Innsbruck, Austria

REFERENCES:
- [Derived] Dammerer D, Liebensteiner M, Rochau H, Uprimny C, Smekal V, Rosenberger R, Servien E. Influence of the anterior notch in mobile-bearing UKA on patellofemoral radiotracer uptake and clinical outcome. BMC Musculoskelet Disord. 2017 Dec 16;18(1):532. doi: 10.1186/s12891-017-1885-6. PMID 29246134